CLINICAL TRIAL: NCT07003919
Title: A Phase 3, Double-Blind, Placebo-Controlled, Randomized Study to Assess the Safety of Epicutaneous Immunotherapy With DBV712 250 mcg in 1-through 3-year-old Children With Peanut Allergy
Brief Title: Safety Study of Viaskin® Peanut Patch in Peanut-Allergic Children 1 Through 3 Years of Age (COMFORT Toddlers)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V712-308
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Allergy; Peanut Allergy
Keywords: Peanut hypersensitivity; Epicutaneous Immunotherapy (EPIT); Epicutaneous; Immunotherapy; Viaskin; Nut and Peanut Hypersensitivity; Food Hypersensitivity; Peanut Allergy; Food Allergy; Nut and Peanut Allergy; Safety Study
MeSH Terms: conditions — Hypersensitivity; Peanut Hypersensitivity; Nut and Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DBPC Treatment Period: DBV712 250 mcg (Experimental): Participants will apply DBV712 250 mcg, epicutaneous system (or patch), daily for a period of 6 months.
  Interventions: Combination Product: DBV712 250 mcg
- DBPC Treatment Period: Placebo (Placebo Comparator): Participants will apply DBV712 matching placebo epicutaneous system (or patch), daily for a period of 6 months.
  Interventions: Combination Product: Placebo
- Optional Open-Label Extension-Period: DBV712 250 mcg (Experimental): The 6-month DBPC period will be followed by an optional open-label extension (OLE) period during which eligible participants will receive DBV712 250 mcg for a duration of 18 months (representing 24 months of active treatment for those participants initially randomized to DBV712 250 mcg and 18 months of active treatment for those participants that were initially randomized to placebo).
  Interventions: Combination Product: DBV712 250 mcg

INTERVENTIONS:
Combination Product: DBV712 250 mcg — DBV712 250 mcg epicutaneous system.
  Other Names: Viaskin® Peanut Patch
  Arms: DBPC Treatment Period: DBV712 250 mcg; Optional Open-Label Extension-Period: DBV712 250 mcg
Combination Product: Placebo — DBV712 matching placebo epicutaneous system.
  Arms: DBPC Treatment Period: Placebo

SUMMARY:
The primary objective of this study is to assess the 6-month safety of DBV712 250 micrograms (mcg) in subjects 1 through 3 years of age with peanut allergy.

DETAILED DESCRIPTION:
This is a Phase 3 randomized double-blind, placebo-controlled (DBPC) study of 6-months duration to assess the safety of DBV712 250 mcg in subjects 1 through 3 years of age with peanut allergy. Participants who complete the 6-month DBPC period will be eligible to enter an optional 18-month open-label extension (OLE).

The overall maximum study duration for each participant will be approximately 112 weeks: Screening Period of 6-weeks, DBPC Treatment Period of 26-weeks, Open-label Period of 78-weeks and Follow-up Period of 2-weeks.

For participation eligibility, please refer to eligibility criteria section.

Randomization of eligible participants will occur in a 3:1 ratio to DBV712 250 mcg (active treatment) or placebo, respectively.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 1 through 3 years at Visit 1 (screening).
* Physician-diagnosed peanut allergy and following a strict peanut-free diet
* Peanut-specific IgE > 0.7 kUA/L.
* A positive peanut SPT with the largest wheal diameter of ≥ 6 mm at Visit 1 (screening).
* An ED ≤ 300 mg peanut protein at screening double-blind placebo-controlled food challenge (DBPCFC).

Key Exclusion Criteria:

* Peanut allergic subjects presenting a medical history of severe anaphylaxis to peanut.
* Severe generalized dermatologic disease involving the proposed treatment application area (interscapular region).
* Current immunotherapy for any allergen (including food allergy, allergic rhinitis and/or insect allergy).
* History of any immunotherapy for peanut allergy, including Epicutaneous immunotherapy (EPIT), oral immunotherapy (OIT), sublingual immunotherapy (SLIT).
* Treatment with any monoclonal antibody or biologic immunomodulatory therapy within 6 months prior to Visit 1.
* Uncontrolled persistent asthma.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
DBPC Treatment Period: Adverse Events (AEs), Treatment-Emergent Adverse Events (TEAEs), and Serious Adverse Events (SAEs) | Through DBPC Treatment Period, 6 months

OTHER OUTCOMES:
Concentration of peanut-specific IgE (kUA/L) at baseline and month 6. | Month 6
Concentration of peanut-specific IgG4 (mg/L) at baseline and month 6. | Month 6
DBPC Treatment Period: Change from baseline in peanut Skin Prick Test (SPT) mean wheal diameters | Month 6

CONTACTS AND LOCATIONS:
Locations (89):
- United States (54):
  - AllerVie Clinical Research, Birmingham, Alabama
  - University of Alabama at Birmingham Pediatric Primary Care Clinic, Birmingham, Alabama
  - Modena Allergy & Asthma, Scottsdale, Arizona
  - University of Arizona Asthma and Airway Disease Research Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Modena Allergy & Asthma, La Jolla, California
  - Modena Allergy and Asthma, Long Beach, California
  - UCLA Health Westwood Pediatrics, Los Angeles, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Allergy & Asthma Medical Group and Research Center, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Asthma & Allergy Associates, Colorado Springs, Colorado
  - Children's National - Main Hospital, Washington D.C., District of Columbia
  - University of South Florida Children's Research Institute, St. Petersburg, Florida
  - Allergy, Asthma & Immunology Associates of Tampa Bay, Tampa, Florida
  - Emory University - Children's Healthcare of Atlanta, Inc., Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago Medicine Comer Children's Hospital, Chicago, Illinois
  - Sneeze, Wheeze and Itch Associated, LLC, Normal, Illinois
  - Deaconess Clinic - Downtown Evansville, Evansville, Indiana
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - The University of Kansas Health System - Main Campus, Medical Pavilion, Kansas City, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - MassGeneral Hospital for Children, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Regents of the University of Michigan, Ann Arbor, Michigan
  - Allergy and Immunology Associates of Ann Arbor, Ann Arbor, Michigan
  - Allergy and Asthma Research Center of Minnesota, Maplewood, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Weiss Medical, Riverdale, New Jersey
  - Northwell Health Allergy and Immunology at the Irving Goldman Family Care Center, Great Neck, New York
  - NYU Langone Health, New York, New York
  - Equity Medical, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - UNC Hospitals Children's Specialty Clinics in Chapel Hill at Carolina Pointe II, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Texas Children's Hospital, Houston, Texas
  - Gundersen Health System - La Crosse Campus, La Crosse, Wisconsin
  - Children's Wisconsin, The Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Westmead Childrens Hospital, Westmead, New South Wales
  - Queensland Children's Hospital and Health Service, South Brisbane, Queensland
  - Royal Children's Hospital Melbourne, Parkville, Victoria
  - Epworth Healthcare Richmond, Richmond, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- Canada (8):
  - Manitoba Allergy Research, Inc., Winnipeg, Manitoba
  - Halton Pediatric Allergy, Burlington, Ontario
  - Hamilton Allergy, Hamilton, Ontario
  - McMaster University Medical Center, Hamilton, Ontario
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - Sick Kids, The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Clinique Specialisee en Allergie de la Capitale, Québec, Quebec
- France (6):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hospices Civils of Lyon, Hôpital Femme Mère Enfant, Bron
  - Centre Hospitalier Régional Universitaire de Lille Hôpital Jeanne de Flandre, Lille
  - Centre Hospitalier Universitaire Montpellier, Montpellier
  - Assistance Publique Hôpitaux de Paris Hôpital Robert Debré, Paris
  - Centre Hospitalier Régional Universitaire de Nancy, Vandœuvre-lès-Nancy
- Ireland (2):
  - Cork University Hospital, Cork
  - Royal College of Surgeons in Ireland. Children's Health Ireland (CHI) at Crumlin, Dublin
- Netherlands (2):
  - Erasmus MC Sophia Children's Hospital, Rotterdam
  - University Medical Center Utrecht (UMCU), Utrecht
- Spain (5):
  - Institut de Recerca Sant Joan de Déu., Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario Ramón y Caja, Madrid
  - Hospital Regional Universitario de Málaga, Hospital Materno Infantil, Málaga
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
- United Kingdom (7):
  - Royal Hospital for Children, Glasgow
  - University Hospitals of Leicester NHS Trust, Leicester
  - Guy's and Saint Thomas' NHS Foundation Trust St Thomas' Hospital, London
  - Allergy Centre of Excellence, London
  - Royal Manchester Children's Hospital, Manchester University NHS Foundation Trust, Manchester
  - Sheffield Children's NHS Foundation Trust Sheffield Children's Hospital, Sheffield
  - University Hospital Southampton NHS Foundation Trust Southampton Children's Hospital, Southampton